CLINICAL TRIAL: NCT06353802
Title: Correlation Between Chronic Non-specific Neck Pain and Lumbar Reposition Sense: a Correlative Study
Brief Title: Relationship Between Chronic Non-Specific Neck Pain And Lumbar Reposition Sense
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammed Hesham Abdelaziz, Principal Investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P.T.REC/012/004963
Record Dates: First submitted 2024-03-28; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Chronic Non-specific Neck Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- group 1 (Other): Participants will be measured using iPhone® Inclinometer Application. The measurement app level, a measuring tool, was utilised with the iPhone® 10 (Apple Inc., California, USA). A free application that is built into the iPhone®, The measurement app level shows the numerical size in a manner similar to a digital inclinometer. The programme shows the angle measured using a digital display and the accelerometer included into the iPhone®. Degrees (°) were used as the measurement unit.
  Interventions: Diagnostic Test: Chronic non-specific neck pain and lumbar reposition sense

INTERVENTIONS:
Diagnostic Test: Chronic non-specific neck pain and lumbar reposition sense — In order to evaluate the lumbar joint repositioning error using the Joint Positioning Sense, the following guidelines were followed: (I) The participants were to stand with their arms at their sides, their feet externally rotated (about 20 degrees).
  (II) With the feet flat on the floor and the arms resting on the front of the thighs, the person was seated in a height-adjustable seat that measured the length of the shank. (III) With a belt fastened, the iPhone® was positioned upright just above the iliac crest, (IV) the inclination of the inclinometer was 0°; (V) The inclinometer's 0° point was set as the initial position. (VI) The individual was passively guided by the assessor to a 30° flexion within the range of 0 to 30°; (VII) the subject was to memorize this position for 10 s; (VIII) the subject actively returned to the initial position. (IX) Subsequently, the participant was required to actively replicate the position three times.

SUMMARY:
to investigate the correlation between chronic non-specific neck pain and lumbar reposition sense.

DETAILED DESCRIPTION:
Around 67% of people on the planet may at some point in their lives experience chronic, non-specific neck pain. People who have chronic pain frequently need medical services and medications for pain treatment, and there is a link between their functional limitations and disabilities.

Cervical pain without a recognized clinical reason for the complaints is classified as chronic non-specific neck pain. Some symptoms include weakening in the neck muscles and reduced mobility of the cervical spine.

"Pain perceived anywhere in the posterior region of the cervical spine, from the superior nuchal line to the first thoracic spinous process" is how the International Association for the Study of Pain (IASP) characterized chronic non-specific neck pain.

Individuals who experience unilateral or central neck discomfort are said to have persistent non-specific neck pain. There will be restricted range of motion in the neck, which frequently re-creates the symptoms; referred shoulder girdle or upper extremity pain may also be felt. Patients may also get cervicogenic headaches (CGH).

Spine position, stability, and movement are all governed by motor control, which results from the ongoing interaction of sensory inputs, such as proprioception, on different neural system levels, and motor outputs to effectors, such as paraspinal muscles.

The capacity to precisely position the trunk at predefined points along the sagittal plane's range of motion is known as trunk position sense. Trunk repositioning protocols may be a valuable tool for measuring trunk control since they demand that participants precisely move and control the flexing trunk.

The most popular criterion for assessing proprioceptive senses is joint repositioning errors. By first generating a target angle or joint location using position or movement sensors, then having the subject represent that place, the test examines the discrepancy between the initial target location and the location realised by the subject.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients,18-50 years old
2. Neck pain continued for at least the last 12 weeks
3. Normal Body mass index ranged from 18.5 to 24.9

Exclusion Criteria:

1. Radiated neck pain
2. Neck pain associated with vertigo
3. A history of surgery on the lower limbs or back
4. Back or lower extremity trauma within the last three months.
5. neurological or vestibular disorders
6. Diagnosed psychological disorders
7. Vertebral fractures
8. Metal spine implants
9. Tumors
10. Diagnosed metabolic diseases
11. Using medications that could have an impact on balance in the 24 hours before to the study
12. Previous neck surgery
13. Red flags (night pain, severe muscle spasms, sudden loss of weight)
14. Physiotherapeutic treatment continued in the last 3 months
15. Pregnancy, including six months postpartum
16. A diagnosed psychiatric disorder or severe cognitive impairment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Correlation Between Chronic Non-Specific Neck Pain And Lumbar Reposition Sense Using iPhone inclinometer app | one month
  using the iPhone inclinometer app to asses the lumbar reposition error measures with degrees and it's correlation to cervical non-specific neck pain using visual analogue scale ranging from 1 to 10

CONTACTS AND LOCATIONS:
Locations (1):
- Physical Therapy College Cairo University, Giza, Egypt